CLINICAL TRIAL: NCT00029237
Title: Alternative Stress Management Approaches in HIV Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: R01AT000331 (NIH)
Record Dates: First submitted 2002-01-09; First posted 2002-01-10 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: HIV Infections
Keywords: Behavioral intervention; Psychoneuroimmunology; Complementary therapy; Stress and coping; complementary therapies
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Behavioral: Cognitive-behavioral relaxation (Positively Living)
Behavioral: Spiritual growth group
Behavioral: Focused Tai Chi

SUMMARY:
The overall purpose of the proposed study is to determine whether three short-term stress management interventions along with booster strategies will improve and sustain improvements in psychosocial functioning, quality of life, and somatic health among persons with varying stages of HIV disease. The 10-week group interventions are designed to reduce perceived stress and increase coping effectiveness and include cognitive-behavioral stress management focused on positively living (+LIVE), focused Tai Chi (TCHI) training, and spiritual growth groups (SPRT). Effects of the interventions will be evaluated immediately upon completion of the group training and at 6 months and 12 months following stress management training.

DETAILED DESCRIPTION:
The overall purpose of the proposed study is to determine whether three short-term stress management interventions along with booster strategies will improve and sustain improvements in the domains of psychosocial functioning, quality of life, and somatic health among persons with varying stages of HIV disease. These three outcome domains, along with neuroendocrine mediation, will be measured by multiple indicators derived from the psychoneuroimmunology (PNI)paradigm. The interventions are designed to reduce perceived stress and increase coping effectiveness and include cognitive-behavioral stress management focused on positively living (+LIVE), focused Tai Chi (TCHI) training, and spiritual growth groups (SPRT). The primary aim of this randomized clinical trial is to compare the +LIVE, TCHI, and SPRT interventions to each other and to standard care received by a control group of wait-listed participants (WAIT) for effects on psychosocial functioning (perceived stress, coping patterns, social support, psychological distress), quality of life (including spiritual well-being), neuroendocrine mediation (cortisol, DHEA levels), and somatic health (disease progression, HIV-specific health status, immune status).

ELIGIBILITY:
Inclusion Criteria:

* Aware of HIV-infected diagnosis

Exclusion Criteria:

* Current psychoactive drug use
* Severe and unstable psychiatric diagnosis
* Major cognitive dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392
Dates: Start 2000-09; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States